CLINICAL TRIAL: NCT06286085
Title: A Comparison of Diagnostic Testing Modalities in the Assessment of Asthma
Acronym: MODELS
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 337788
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: lung function; impulse oscillometry
MeSH Terms: conditions — Asthma | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Lung function tests — Pulmonary function tests

SUMMARY:
This study aims to assess the concordance of international asthma guidelines in the diagnosis of asthma and explore the presence of airways disease using additional non-guideline physiologic criteria, such as IOS (impulse osciollometry), not included in the guidelines, but available in the Portsmouth lung function service.

DETAILED DESCRIPTION:
Asthma is a widespread condition that affects millions of people worldwide. It is characterized by symptoms such as difficulty breathing, coughing, and wheezing. Diagnosing asthma involves identifying certain indicators like airflow obstruction, airway sensitivity, and inflammation. However, different international guidelines, including those from organizations such as NICE (National Institute for Health and Care Excellence), GINA (Global Initiative for Asthma), and BTS (British Thoracic Society)/SIGN (Scottish Intercollegiate Guidelines Network), have varying criteria for diagnosis. This can lead to inconsistencies in identifying patients with asthma.

This study aims to evaluate the effectiveness of different diagnostic approaches, including impulse oscillometry (IOS), in diagnosing asthma. IOS is a simple and non-invasive test that measures lung function. It has the potential to enhance the accuracy and ease of asthma diagnosis. Despite its promise, current research on the role of IOS in diagnosing asthma in adults is limited.

To address these gaps in knowledge, the study will examine the data of patients attending the severe asthma service at Queen Alexandra Hospital in Portsmouth. With an "opt-out" consent process, routine outpatient lung function data will be analysed, paying special attention to the usefulness of IOS compared to other lung function indices in diagnosing asthma.

By conducting this study, the aim is to contribute valuable insights to the field of asthma diagnosis. The study findings may help refine the methodology of diagnosing asthma and potentially expand the diagnostic toolkit to include IOS. This could improve the precision and ease of managing asthma, leading to better outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient will meet all the following criteria to be considered eligible for the study:

  * Aged 18 years or over.
  * All patients who have attended full asthma workups from November 2021 till date
  * Willing and able to consent to use their data in this study (opt-out form or e-consent).
  * Patients referred to the Portsmouth asthma service for diagnosis and further management of presumed asthma. Comorbidities are common in asthma, thus patients with co-existing conditions such as obesity, bronchiectasis or COPD will be included.

Exclusion Criteria:

* The participant may not enter the study if either of the following apply:

  * Unable to comprehend the study and provide informed consent, e.g., insufficient command of English in the absence of someone who can adequately interpret.
  * Patients with other primary respiratory conditions, such as ILD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients referred for specialist review from primary care and needing specialist review after emergency admission. This research will utilise historical and contemporary data from pulmonary function tests performed during the asthma workup at the Queen Alexandra Hospital, Portsmouth. The tests will include Fractional Exhaled Nitric Oxide (FeNO), Skin prick tests, Impulse Oscillometry, Spirometry, Gas transfer, lung volumes and Bronchodilator reversibility.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2027-05-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
International asthma guidelines scores | during study analysis 4 weeks after recruitment
  To assess the levels of concordance among international asthma guidelines for the diagnosis of asthma in patients referred to a secondary/tertiary care asthma service.
non-guideline physiologic criteria numbers | during study analysis 4 weeks after recruitment
  Assess the presence or absence of airway disease by the non-guideline physiologic criteria with those fulfilling (or not) the diagnostic criteria for asthma according to any of the selected guidelines.

SECONDARY OUTCOMES:
non-guideline physiologic criteria for asthma. | during study analysis 4 weeks after recruitment
  Compare the clinical characteristics of patients stratified by the presence or absence of guideline and non-guideline physiologic criteria for asthma.
Comparison of the diagnostic outcomes of each guideline with a "reference standard". | during study analysis 4 weeks after recruitment
  Assess the sensitivity of each guideline in the diagnosis of airway disease by comparing the diagnostic outcomes of each guideline with a "reference standard".

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Chauhan, Principal Investigator — Portsmouth University Hospital Trust
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared.